CLINICAL TRIAL: NCT04819126
Title: Nintendo Wii Virtual Reality Application In Older People With Alzheimer's Dementia
Brief Title: Nintendo Wii Virtual Reality Application In Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meral SERTEL, Kırıkkale University, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Karamanoğlu Mehmet Bey U; Kırıkkale University (Other: Kırıkkale University)
Record Dates: First submitted 2021-03-10; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Age-Related Memory Disorders
Keywords: Alzheimer's Dementia; Muscle strength; Fall; Virtual reality
MeSH Terms: conditions — Memory Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nintendo Wii Virtual Reality Application In Older People With Alzheimer's Dementia (Experimental): The study included a total of 32 volunteers between the ages of 65-80, who stayed in Karaman Ahmet Mete Nursing Home, Elderly Care and Rehabilitation Center, with mild or moderate Alzheimer's dementia diagnosed by a neurologist. As a result of the power analysis, it was calculated that at least 16 individuals could be included in each group (at least 32 individuals in total). Randomization was performed by the sealed-envelope method. According to this method, 4 females and 12 males were determined to be in the control group, while 5 females and 11 males were determined to be in the training group.
  The evaluation was completed before the intervention. The same evaluation was conducted after 6 weeks.
  The training group was trained with games from different categories such as balance and aerobic exercises with a Nintendo Wii virtual reality device 2 times a week for a period of 6 weeks, with 1 session lasting for 30 minutes, and each patient was trained with the same games.
  Interventions: Other: Nintendo Wii Virtual Reality Application
- Older People With Alzheimer's Dementia (No Intervention): In the control group, no application was performed during this period, and routine medical treatments were continued. The training group was evaluated before and after the training, while the control group was re-evaluated at the end of the 6th week after the first evaluation. After the study was completed, the volunteers from the control group were also given training.

INTERVENTIONS:
Other: Nintendo Wii Virtual Reality Application — The training group was trained with games from different categories such as balance and aerobic exercises with a Nintendo Wii virtual reality device 2 times a week for a period of 6 weeks, with 1 session lasting for 30 minutes.
  Arms: Nintendo Wii Virtual Reality Application In Older People With Alzheimer's Dementia

SUMMARY:
•This study was planned to investigate the effects of the Nintendo Wii virtual reality application on muscle strength and fall risk in individuals with AD.

The aim of the present study is to investigate the effect of the virtual reality application on muscle strength and fall in individuals with Alzheimer' Dementia (AD).

DETAILED DESCRIPTION:
Purpose: This study was planned to investigate the effects of the Nintendo Wii virtual reality application on muscle strength and fall risk in individuals with AD.

Method: The study included a total of 32 volunteers between the ages of 65-80, with mild or moderate AD diagnosed. These individuals were divided into 2 groups as a training group and control group. The training group was trained with games from different categories such as balance and aerobic exercises with a Nintendo Wii virtual reality device 2 times a week for a period of 6 weeks, with 1 session lasting for 30 minutes. Mini-Mental State Test, Knee Extension Muscle Strength, Timed Up and Go Test, Tinetti Falls Efficacy Scale results of individuals were recorded in the evaluation.

ELIGIBILITY:
Inclusion Criteria:

* included volunteers between the ages of 65-80 with mild or moderate AD diagnosis,
* who did not have any difficulty or problems in communicating,
* who did not have any neurological diseases that disrupt balance and coordination such as a cerebrovascular event, Parkinson's disease, Multiple Sclerosis, and neurological disorder,
* who obtained a score of 18 - 24 points in the Mini-Mental State Test (MMST)

Exclusion Criteria:

* Patients diagnosed with rapidly progressing dementia (infection, vascular, hematologic diseases),
* Those who could not be contacted during the follow-up period or who did not participate in the training session, those who experienced cardiac and cerebrovascular events, endocrine disorders, fluid-electrolyte imbalance and infection,
* Those with malignancy and those who received chemotherapy and radiotherapy that causes malignancy, delirium or depression and malignant sensory loss (those with the Semmes-Weinstein monofilament thickness of 4.56 and above),
* Those with a lower or upper extremity amputation at any level

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Age :mean or median age | period of 6 weeks
  Age, Categorical:
  >=65 years
Body Mass Index | period of 6 weeks
  BMI was recorded in kg/m^2.
Sex/Gender | period of 6 weeks
  Sex: Female, Male

SECONDARY OUTCOMES:
The Mini-Mental State Test for Cognitive status | period of 6 weeks
  According to the MMST, 24-30 points were considered as normal cognitive levels, 18-23 points were considered as mild cognitive disorders, and 0-17 points were considered as severe cognitive disorders

CONTACTS AND LOCATIONS:
Overall Officials: Konya Karaman Ahmet Mete Nursing Home, Principal Investigator — Karaman Ahmet Mete Nursing Home. Konya in Turkey
Locations (1):
- Karaman Ahmet Mete Nursing Home, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT04819126/Prot_SAP_ICF_000.pdf